CLINICAL TRIAL: NCT02957695
Title: Neurofeedback in Patients With Frontal Brain Lesions: Randomised Controlled Double-blind Trial
Brief Title: Neurofeedback in Patients With Frontal Brain Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PD Dr. med. Margret Hund-Georgiadis (Other)
Collaborators: Rehab Basel (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Margret Hund-Georgiadis, PD Dr. med., Rehab Basel
Organization: Rehab Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EKNZ 2015-105
Record Dates: First submitted 2016-03-13; First posted 2016-11-08 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Brain Lesion
Keywords: frontal brain lesions; neurofeedback; cognitive functions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Control Intervention: Placebo-Neurofeedback, 20 sessions
  Interventions: Device: Placebo-Neurofeedback
- Intervention group (Active Comparator): Experimental Intervention: Active-Neurofeedback, 20 sessions
  Interventions: Device: Active-Neurofeedback

INTERVENTIONS:
Device: Placebo-Neurofeedback — The Intervention used for the control-group consists of a sham-neurofeedback, which is based on a previous eeg-recording and doesn't respond to the actual brain activity. The fact, that it is not a real neurofeedback, cannot be recognized by the patient nor the trainer because the eeg recording is not visible and the program reacts to muscle contractions (where feedback reactions would be expected) but not to brain activity.
  Arms: Control group
Device: Active-Neurofeedback — The neurofeedback-method used in our study is called "infra-low frequency neurofeedback Training", developed by S. and S. Othmer. NeuroAmpII® is the device and Cygnet® the corresponding Software used for this method, both are approved as an active medicinal device (CE-marked) in the European Union and in USA (www.eeginfo.com). The device and the Software are produced by the Company BEE Medic GmbH, Kirchberg, CH.
  Arms: Intervention group

SUMMARY:
In this randomized double-blind controlled study we would like to test the benefit of neurofeedback for the recovery of patients with frontal brain injury during an early stage of neurorehabilitation.

DETAILED DESCRIPTION:
Aim of the study: Patients with a frontal brain lesion often suffer from deficits in brain functions like attention, concentration, planning, impulse control and emotional stability. In this study the investigators would like to test, whether neurofeedback as a non-medication option can help to improve these cognitive functions. Neurofeedback is a method for optimization and stabilization of the brain activity. The brain continuously gets computer-based information about its state. This information is used by the brain for self-regulation. Because neurofeedback is a process based on learning, the positive effects can be integrated into the daily life and seem to persist also after the training stopped. From the literature, several studies have shown promising results of neurofeedback therapy in patients with brain injuries, but no study so far fulfills the scientific criteria which proves a benefit. Methods: The selection of potential study participants is made by the senior or chief physician. Totally, we include 20 patients with a newly acquired frontal brain lesion. 10 patients receive normal neurofeedback training and 10 patients receive a placebo-neurofeedback in a randomized, double blinded manner. In total, 20 neurofeedback sessions are conducted. At the beginning, after 10 sessions and at the end of the intervention time, a neuropsychological assessment is performed to test the main cognitive functions of the frontal brain. Data analysis: The performance in the neuropsychological testing is the primary outcome. We expect that all participants will gain performance during the course of the study due to natural brain recovery, so that we will focus on the difference of the improvements between the two groups (neurofeedback and placebo-group).

ELIGIBILITY:
Inclusion criteria:

* Middle to severe frontal or frontotemporal brain injury due to accident, bleeding or ischemia, assessed by the Initial Glascow-Coma-Scale from 3 to 12.
* Time between the injury and inclusion into the study should be 1-6 months
* The participants must be able to perform simple neuropsychologic tests including sufficient vigilance and motor function for pressing a button.
* There is no age limitation. The patients who are hospitalized in the REHAB for a initial rehabilitation have a minimum age of 18 years.
* signed consent form

Exclusion criteria:

* therapy-resistant symptomatic epilepsy
* severe cognitive deficits, which do not allow understanding of the required neuropsychological tests, e.g. sensory aphasia.
* preexisting dementia
* progressive cerebral diseases e.g. multiple sclerosis, brain tumor
* schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in frontal brain function assessed by FAB (Frontal assessment battery) scale | Assessments are made before intervention, after 4 weeks of intervention and after 8 weeks of intervention
  1. Change in the FAB scale (point score) assessed before, after 4 weeks of intervention and after 8 weeks of intervention
Change in frontal brain function assessed by Alertness Test | Assessments are made before intervention, after 4 weeks of intervention and after 8 weeks of intervention
  Change in the Alertness Test (T-values) assessed before, after 4 weeks of intervention and after 8 weeks of intervention
Change in frontal brain function assessed by the GoNogo-Test | Assessments are made before intervention, after 4 weeks of intervention and after 8 weeks of intervention
  Change in the GoNogo-Test (T-values) assessed before, after 4 weeks of intervention and after 8 weeks of intervention
Change in frontal brain function assessed by the Emotion recognition Test | Assessments are made before intervention, after 4 weeks of intervention and after 8 weeks of intervention
  Change in the Emotion recognition Test (T-values) assessed before, after 4 weeks of intervention and after 8 weeks of intervention

SECONDARY OUTCOMES:
Change in behaviour assessed by the Frontal Systems Behavioral Scale (FrSBe) | Assessments are made before intervention, after 4 weeks of intervention and after 8 weeks of intervention
  FrSBe is a questionnaire to assess behaviour as an important frontal brain function. This questionnaire is filled out by the responsible nurse and as a self-rating form by the patient himself. The improvement in behaviour measured by the questionnaire (T-values) assessed before, after 4 weeks and after 8 weeks of Intervention is a secondary outcome.
Change in quantitative eeg z-scores of coherence and relative power | Assessment is made before and after 8 weeks of intervention
  Difference in z-scores of quantitative eeg measured before and after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Margret Hund-Georgiadis, MD, PD, Principal Investigator — REHAB Basel, Switzerland
Locations (1):
- Rehab Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benke T, Karner E, Delazer M. FAB-D: German version of the Frontal Assessment Battery. J Neurol. 2013 Aug;260(8):2066-72. doi: 10.1007/s00415-013-6929-8. Epub 2013 May 7. PMID 23649609
- [Background] Gevensleben H, Holl B, Albrecht B, Vogel C, Schlamp D, Kratz O, Studer P, Rothenberger A, Moll GH, Heinrich H. Is neurofeedback an efficacious treatment for ADHD? A randomised controlled clinical trial. J Child Psychol Psychiatry. 2009 Jul;50(7):780-9. doi: 10.1111/j.1469-7610.2008.02033.x. Epub 2009 Jan 12. PMID 19207632
- [Background] Levesque J, Beauregard M, Mensour B. Effect of neurofeedback training on the neural substrates of selective attention in children with attention-deficit/hyperactivity disorder: a functional magnetic resonance imaging study. Neurosci Lett. 2006 Feb 20;394(3):216-21. doi: 10.1016/j.neulet.2005.10.100. Epub 2005 Dec 15. PMID 16343769
- [Background] May G, Benson R, Balon R, Boutros N. Neurofeedback and traumatic brain injury: a literature review. Ann Clin Psychiatry. 2013 Nov;25(4):289-96. PMID 24199220
- [Background] Steiner NJ, Sheldrick RC, Gotthelf D, Perrin EC. Computer-based attention training in the schools for children with attention deficit/hyperactivity disorder: a preliminary trial. Clin Pediatr (Phila). 2011 Jul;50(7):615-22. doi: 10.1177/0009922810397887. Epub 2011 May 10. PMID 21561933
- [Background] Wangler S, Gevensleben H, Albrecht B, Studer P, Rothenberger A, Moll GH, Heinrich H. Neurofeedback in children with ADHD: specific event-related potential findings of a randomized controlled trial. Clin Neurophysiol. 2011 May;122(5):942-50. doi: 10.1016/j.clinph.2010.06.036. Epub 2010 Sep 16. PMID 20843737
- [Derived] Annaheim C, Hug K, Stumm C, Messerli M, Simon Y, Hund-Georgiadis M. Neurofeedback in patients with frontal brain lesions: A randomized, controlled double-blind trial. Front Hum Neurosci. 2022 Sep 15;16:979723. doi: 10.3389/fnhum.2022.979723. eCollection 2022. PMID 36188178